CLINICAL TRIAL: NCT05411822
Title: Understanding Circadian Responses to Light in Persons With Mild Cognitive Impairment and Alzheimer's Disease
Brief Title: Understanding Circadian Responses to Light in Persons With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 21-0400; R21AG070713 (NIH)
Record Dates: First submitted 2022-06-02; First posted 2022-06-09 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Mild Cognitive Impairment (Experimental): Every participant experienced all 5 conditions:
  Blue light (λmax = 451 nm) on axis and off axis.
  Green light (λmax = 522 nm) on and off axis
  Dim-light control condition (< 5 lux at the eye) for 30 min
  each narrowband source will have distinct lighting distribution patterns but calibrated to deliver the same targeted levels of circadian light (CLA) and circadian stimulus (CS) at the eye.
  Interventions: Device: Lighting Intervention Blue light; Device: Lighting Intervention Green light; Other: Dim-light control condition

INTERVENTIONS:
Device: Lighting Intervention Blue light — Custom made lighting fixture that will deliver the blue lighting intervention. Blue light (λmax = 451 nm) on axis and off axis.
Device: Lighting Intervention Green light — Custom made lighting fixture that will deliver the green lighting intervention. Green light (λmax = 522 nm) on and off axis
Other: Dim-light control condition — (< 5 lux at the eye) for 30 min

SUMMARY:
The purpose of this research study is to investigate the relationship between light, the thickness of the pigment at the back of your eye, melatonin levels, and memory. The study will investigate whether changing light distribution pattern from "on-axis"' (i.e., directed along the eye's visual axis to the fovea) to "off-axis" (i.e., directed on the periphery of the eye's visual axis) impact melatonin suppression in 24 mild cognitive impairment participants and 24 healthy, age-matched controls.

DETAILED DESCRIPTION:
Eligible enrolled subjects will be exposed to 4 different lighting conditions in addition to one dark control condition. There will be 5 study session and each one will last for 90 minutes and will be separated by one week. Subjects will collect 3 saliva samples, each one 30 minutes apart for melatonin levels during each study session.

ELIGIBILITY:
Inclusion Criteria:

* mild cognitive impairment
* age matched healthy control
* macular pigment density either < 0.3 or > 0.5

Exclusion Criteria:

* extensive brain vascular disease
* Parkinson's disease
* bipolar disorder
* seasonal depression
* diabetes
* high blood pressure
* obstructing cataracts
* macular degeneration
* diabetic retinopathy
* use of melatonin supplements
* use of beta blockers
* use of sleep medications
* use of antidepressant medication

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, PhD, Principal Investigator — Icahn School of Medicine
Locations (1):
- Light and Health Research Center at Mount Sinai, Menands, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Matched Control: Healthy Age-Matched Control
Period: Overall Study
Arm/Group | Participants With Mild Cognitive Impairment | Matched Control
Started | 17 | 19
Completed | 15 | 18
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Healthy Age-Matched Control: Healthy Age-Matched Control
- Total: Total of all reporting groups
Arm/Group | Participants With Mild Cognitive Impairment | Healthy Age-Matched Control | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (7.4) | 58.7 (7.6) | 58.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 2 | 6 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Melatonin Levels
Description: Saliva samples collected for melatonin levels for the different conditions. Blue light (λmax = 451 nm) on axis and off axis: for each narrowband source, designated on-axis or off-axis, will have distinct lighting distribution patterns but calibrated to deliver the same targeted levels of circadian light (CLA) and circadian stimulus (CS) at the eye.
  Green light (λmax = 522 nm) on and off axis: for each narrowband source, designated on-axis or off-axis, will have distinct lighting distribution patterns but calibrated to deliver the same targeted levels of circadian light (CLA) and circadian stimulus (CS) at the eye.
  Dim-light control condition: (< 5 lux at the eye) for 30 min
Time Frame: post-intervention (60 minutes) on each night of intervention (one night a week for 5 weeks)
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Mild Cognitive Impairment: Participants who have mild cognitive impairment
- Healthy Control: Participants who are healthy.
Arm/Group | Mild Cognitive Impairment | Healthy Control
Number analyzed (Participants) | 13 | 15
pg/mL
  Blue light (λmax = 451 nm) on axis | 0.89 (0.49) | 0.84 (0.51)
  Blue light (λmax = 451 nm) off axis | 0.9 (0.46) | 0.68 (0.21)
  Green light (λmax = 522 nm) on axis | 0.73 (0.14) | 0.73 (0.3)
  Green light (λmax = 522 nm) off axis | 0.82 (0.39) | 0.79 (0.24)
  Dim Light | 1.53 (0.7) | 1.27 (0.3)

ADVERSE EVENTS:
Time Frame: 60 minutes of intervention over 1 day per week for 5 weeks.
Description: Adverse events reporting by comparing conditions. All participants received all conditions.
Groups:
- Mild Cognitive Impairment - Lighting Intervention Blue - On Axis; Healthy Control - Lighting Intervention Blue - On Axis: Blue light (λmax = 451 nm) on axis
  for each narrowband source, designated on-axis, will have distinct lighting distribution patterns but calibrated to deliver the same targeted levels of circadian light (CLA) and circadian stimulus (CS) at the eye.
- Mild Cognitive Impairment - Blue - Off Axis; Healthy Control - Blue - Off Axis: Blue light (λmax = 451 nm)
  for each narrowband source, designated off-axis, will have distinct lighting distribution patterns but calibrated to deliver the same targeted levels of circadian light (CLA) and circadian stimulus (CS) at the eye.
- Mild Cognitive Impairment - Lighting Intervention Green - On Axis; Health Control - Lighting Intervention Green - On Axis: Green light (λmax = 522 nm) on and off axis
  for each narrowband source, designated on-axis, will have distinct lighting distribution patterns but calibrated to deliver the same targeted levels of circadian light (CLA) and circadian stimulus (CS) at the eye.
- Mild Cognitive Impairment - Green - Off Axis; Healthy Control - Green - Off Axis: Green light (λmax = 522 nm)
  for each narrowband source, designated off-axis, will have distinct lighting distribution patterns but calibrated to deliver the same targeted levels of circadian light (CLA) and circadian stimulus (CS) at the eye.
- Mild Cognitive Impairment - Dim Light; Health Control Dim Light: Dim-light control condition
  (< 5 lux at the eye) for 30 min
Arm/Group | Mild Cognitive Impairment - Lighting Intervention Blue - On Axis | Mild Cognitive Impairment - Blue - Off Axis | Mild Cognitive Impairment - Lighting Intervention Green - On Axis | Mild Cognitive Impairment - Green - Off Axis | Mild Cognitive Impairment - Dim Light | Healthy Control - Lighting Intervention Blue - On Axis | Healthy Control - Blue - Off Axis | Health Control - Lighting Intervention Green - On Axis | Healthy Control - Green - Off Axis | Health Control Dim Light
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13 | 0/13 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13 | 0/13 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13 | 0/13 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT05411822/Prot_SAP_000.pdf